CLINICAL TRIAL: NCT00988663
Title: Memantine Augmentation of Electroconvulsive Therapy in Patients With Major Depression
Brief Title: The Impact of Memantine on Electroconvulsive Therapy (ECT): Will it Improve Response and Protect Against Cognitive Problems?
Acronym: ECTAug
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI deceased; study did not start.
Sponsor: Jerrry L Lewis (Other)
Responsible Party: Sponsor-Investigator, Jerrry L Lewis, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Memantine ECT trial
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Major Depressive Disorder
Keywords: electroconvulsive therapy; memantine; cognitive function; memory
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine arm (Active Comparator): Patient receiving ECT and Memantine
  Interventions: Drug: memantine
- placebo (Placebo Comparator): 25 patients receiving ECT will will receive placebo
  Interventions: Drug: memantine; Drug: Placebo

INTERVENTIONS:
Drug: memantine — patient will receive 5mg daily for 7day then 10 mgm daily
  Other Names: Namenda
Drug: Placebo — will give placebo that looks like memantine
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether memantine will enhance the therapeutic of effect on depression and prevent memory and other cognitive problems caused by ECT.

DETAILED DESCRIPTION:
Patients will be assigned randomly either to a treatment group or a placebo groups. All patients in both groups will be receiving standard ECT. The treatment group will receive memantine. All patients will be given a battery of cognitive tests and test of depression before ECT treatments start, after the 6th ECT treatment and after the completions of ECT. An analysis will be performed to see if memantine causes any impact on the response to ECT and prevents memory and cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for Major Depressive disorder

Exclusion Criteria:

* Neurological disease
* Mental retardation
* Seizure disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Assessment of whether Memantine protects memory and cognitive impairment caused by ECT. | 6 to 8 weeks

SECONDARY OUTCOMES:
Whether memantine will improve response of Depression to Electroconvulsive therapy. | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jerry L Lewis, MD, Principal Investigator — University of Iowa Hospitals and Clinic
Locations (1):
- University of Iowa hosptitals and clinic, Iowa City, Iowa, United States